CLINICAL TRIAL: NCT00366808
Title: Mechanical vs. Alcohol Separation of the Corneal Epithelium During Surface Ablation Refractive Procedures
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: MRC-06-003
Record Dates: First submitted 2006-08-17; First posted 2006-08-21 (Estimated); Last update posted 2018-06-14 (Actual); Status verified 2006-07

CONDITIONS: Keratomileusis, Laser In Situ

INTERVENTIONS:
Procedure: LASIK surgery

SUMMARY:
A recent survey of trends among the members of the American Society of Cataract and Refractive Surgery determined that laser in situ keratomileusis (LASIK) is the leading surgical procedure for photorefractive corrections ranging from -0 to 3 diopters (D).1 The same survey, however, showed a clear trend of participating refractive surgeons toward surface ablation. Photorefractive keratectomy (PRK) was the first refractive surgery procedure approved and performed using the excimer laser. Several techniques of epithelial debridement have been tried with PRK-type surgery including mechanical debridement, laser transepithelial ablation, a rotating brush, and alcohol debridement.

The Amadeus II microkeratome (Advanced Medical Optics Inc, Irvine, CA, USA) used for the creation of a LASIK flap has an upgradeable platform that will allow the user to perform mechanical separation of the corneal epithelium before photorefractive treatments. With the use of this device, the corneal epithelium can be separated from the underlying stroma without previous preparation of the corneal surface with alcohol. The separated epithelial sheet can either be removed or replaced on the operated cornea after photoablation. This surgical procedure, which has been called Epi-LASIK, represents an advanced alternative surface ablation photorefractive procedure for the correction of ametropia. The purpose of this study is to evaluate the clinical visual outcomes, healing rates, and patient satisfaction when performing surface ablation procedures using mechanical vs. alcohol separation of the epithelium.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be a candidate for surface ablation procedures in both eyes.
* ≥ 18 years of age or older.
* Myopia ≤ -6.00 D.
* Astigmatism ≤ - 3.00 D.
* Manifest refraction spherical equivalent (MRSE) of -6.00 D.
* Capable of wearing a bandage contact lens.
* Willing and able to comply with scheduled visits and other study procedures.

Exclusion Criteria:

* History of ocular pathology.
* Very large pupils (greater than 8mm diameter, infrared measurement).
* Thin corneas (preoperatively calculated minimal residual bed < 250 um).
* If patient fit into the group of the usual exclusionary criteria (e.g. irregular astigmatism, asymmetric astigmatism, unstable refraction - most of these patients would not typically be considered LASIK candidates under normal circumstances).
* History of previous refractive surgery.
* Corneal irregularities potentially affecting visual acuity: keratoconus, corneal dystrophy, corneal opacities.
* Participation in (or current participation) any investigational drug or device trial within the previous 30 days prior to the start date of this trial.
* Intraocular conventional surgery within the past three months or intraocular laser surgery within one month in the operated eye.
* Use of any systemic or topical drug known to interfere with visual performance.
* Pregnant or nursing mothers and females of childbearing potential not practicing a reliable and medically acceptable method of birth control
* Inability or unwillingness of subjects to give written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10
Dates: Start 2006-02; Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kerry Solomon, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Magill Laser Center, Medical University of South Carolina, Charleston, South Carolina, United States